CLINICAL TRIAL: NCT03655548
Title: Optimization Management Study of Community Urinary Tract Infections Spectrum
Acronym: OPTICUR-EBLSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OPTICUR-EBLSE
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Urinary Tract Infections; Resistant Infection; Community-Acquired Infections; Beta Lactam Resistant Bacterial Infection
MeSH Terms: conditions — Urinary Tract Infections; Community-Acquired Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary tract infections are the second most common community-acquired infections. Even if extended spectrum β-lactamase-producing Enterobacteriaceae (ESBLE) cause fewer urinary tract infections, their proportion is increasing. New recommendations were published by ANSM in 2015, with specific recommendations for infections due to ESBL-producing Enterobacteriaceae. In this study, we wanted to evaluate the effectiveness of a recall of the 2015 recommendations in the form of a table attached to the ECBU report, associated with hygiene recommendations.

Methodology: This prospective, multi-center, non-interventional study was conducted in collaboration with the Labazur laboratory over two 2-month periods, one without modification of the laboratory's practices, the other with the addition of documents on the CBEU report. The primary endpoint was the adequacy of prescriptions to ANSM 2015 recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient who were prescribed by a GP a CBEU during the 2 inclusion periods (from 1/10/2016 to 28/02/2017 with a first period from 01/10/2016 to 30/11/2016 and a second period from 02/01/2016 to 28/02/2017)
* CBEU analyzed by Labazur laboratory
* CBEU positive for a spectrum β-lactamase-producing Enterobacteriaceae (ESBLE)

Exclusion Criteria:

* Children
* Refusal of consent
* CBEU prescribed by a specialist
* patient hospitalised for management of the infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient who were prescribed by a GP a CBEU during the 2 inclusion periods (from 1/10/2016 to 28/02/2017 with a first period from 01/10/2016 to 30/11/2016 and a second period from 02/01/2016 to 28/02/2017)
  * CBEU analyzed by Labazur laboratory
  * CBEU positive for a spectrum β-lactamase-producing Enterobacteriaceae (ESBLE)
  * Ambulatory management of the infection by the GP
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
percentage of adequation to ANSM 2015 guidelines of antibotics prescription for community acquired urinary tract infection before and after CBEU report | One month